CLINICAL TRIAL: NCT00090077
Title: A Phase I, Multicenter, Randomized, Parallel, Double-Blinded Dose Ranging, Placebo-Controlled Study to Compare Antiviral Effect, Safety, Tolerability and Pharmacokinetics of Four Oral Dosage Regimens of GW695634G Monotherapy Versus Placebo Over 10 Days in ART-Naive HIV-1 Infected Adults.
Brief Title: Monotherapy Versus Placebo Over 7 Days-Non-Nucleoside Reverse Transcriptase Inhibitor-Experienced HIV1 Infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN210005
Record Dates: First submitted 2004-08-24; First posted 2004-08-26 (Estimated); Last update posted 2006-02-27 (Estimated); Status verified 2006-02

CONDITIONS: HIV Infections
Keywords: GW695634G; GW695634X; GW678248X; pharmacokinetics; NNRTI; HIV
MeSH Terms: conditions — HIV Infections | interventions — N-(4-(((4-chloro-2-(3-chloro-5-cyanobenzoyl)phenoxy)acetyl)amino)-3-methylphenyl)sulfonylpropanamide

INTERVENTIONS:
Drug: GW695634

SUMMARY:
To investigate safety, tolerability and antiviral activity in Non-nucleoside reverse transcriptase inhibitor (NNRTI)-experienced HIV-1 infected patients

ELIGIBILITY:
Inclusion criteria:

* CD4 cell count greater than or equal to 200 cells/mm3.
* HIV-1 RNA >2000 copies/mL.
* Must have history of NNRTI treatment with subsequent failure and documented evidence of an NNRTI-associated mutation or a phenotype displaying reduced activity to efavirenz, nevirapine or delavirdine.
* Normal resting 12-lead electrocardiogram.

Exclusion criteria:

* Any history of seizure, CNS toxoplasmosis infection, or any CNS (central nervous system) lesion.
* Chronic diarrhea (>3 loose stools/day).
* An active CDC Category C disease (1993), except cutaneous Kaposi's Sarcoma (KS) not requiring systemic therapy during the trial.
* Less than 4 weeks since stopping anti-retroviral therapy (ART) therapy prior to Day 1.
* Any acute laboratory abnormality.
* Positive for HCV antibody or HepBsAG.
* Active infections requiring therapy in the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-04

PRIMARY OUTCOMES:
Safety & tolerability parameters Change from baseline in plasma HIV-1 RNA Change from baseline in CD4+ cell count Plasma GW678248X pharmacokinetic parameters Days 1 & 7

SECONDARY OUTCOMES:
Plasma GW695634X pharmacokinetic parameters on Day 1 and Day 7 Exploratory relationship of pharmacokinetic parameters to changes in virology, immunology and/or safety assessments

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trial, MD, Study Director — GlaxoSmithKline
Locations (18):
- United States (18):
  - GSK Clinical Trials Call Center, Phoenix, Arizona
  - GSK Clinical Trials Call Center, Fountain Valley, California
  - GSK Clinical Trials Call Center, San Francisco, California
  - GSK Clinical Trials Call Center, West Hollywood, California
  - GSK Clinical Trials Call Center, Washington D.C., District of Columbia
  - GSK Clinical Trials Call Center, Fort Lauderdale, Florida
  - GSK Clinical Trials Call Center, Miami, Florida
  - GSK Clinical Trials Call Center, Miami Beach, Florida
  - GSK Clinical Trials Call Center, Orlando, Florida
  - GSK Clinical Trials Call Center, Vero Beach, Florida
  - GSK Clinical Trials Call Center, Atlanta, Georgia
  - GSK Clinical Trials Call Center, Boston, Massachusetts
  - GSK Clinical Trials Call Center, Las Vegas, Nevada
  - GSK Clinical Trials Call Center, New York, New York
  - GSK Clinical Trials Call Center, Charlotte, North Carolina
  - GSK Clinical Trials Call Center, Oklahoma City, Oklahoma
  - GSK Clinical Trials Call Center, Fort Worth, Texas
  - GSK Clinical Trials Call Center, Seattle, Washington